CLINICAL TRIAL: NCT04025944
Title: Real World Study of Chronic Viral Hepatitis
Status: Recruiting | Type: Observational
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, Chief of department of infectious disease, Huashan Hospital
Other Study IDs: KY2019-RWS(CVH)
Record Dates: First submitted 2019-07-07; First posted 2019-07-19 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Hepatitis, Chronic
MeSH Terms: conditions — Hepatitis, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- chronic hepatitis B: No intervention. The clinical data of patients (including demographic information, details of antiviral therapy, imaging and laboratory testings) will be collected and analyzed.
- chronic hepatitis C: No intervention. The clinical data of patients (including demographic information, details of antiviral therapy, imaging and laboratory testings) will be collected and analyzed.

SUMMARY:
This study is aimed to collect and analyze clinical data of patients with chronic viral hepatitis in the real world, to investigate the long-term outcome of these patients and to optimize treatment options based on these data.

DETAILED DESCRIPTION:
Chronic viral hepatitis is defined as infectious liver disease caused by persistent virus infection for more than six months. Sustained viral replication and ongoing liver inflammation can eventually lead to liver fibrosis/cirrhosis or even hepatocellular carcinoma. Chronic viral hepatitis infection causes at least 80% of all liver cancers.

Though chronic viral hepatitis is a major global health concern, there is still a lack of evidence in high quality about the management of chronic viral hepatitis and the long-term outcome of patients. The concept of real-world data and research has been officially introduced into China since 2010. Real-world evidence, based on real-world data, can help practitioners have better understanding of the characteristics of the patients with different treatment strategies.

This study is aimed to collect and analyze clinical data of patients with chronic viral hepatitis in the real world, to investigate the long-term outcome of these patients and to optimize treatment options based on these data.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent of patients.
2. Evidence of persistent virus infection for greater than six months [hepatitis C virus(HCV) RNA positive, hepatitis B surface antigen(HBsAg) or hepatitis B virus(HBV) DNA positive]

Exclusion Criteria:

1. Serious psychiatric history, especially depression.

   * Severe mental illness is defined as major depression or psychosis, suicide attempts, hospitalization due to mental illness or a period of disability due to mental illness.
2. Patients with serious diseases of heart, lung, kidney, brain, blood and other important organs.
3. Patients with malignant tumors (excluding those cured).

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with chronic viral hepatitis.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2019-07-20 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Virologic responses(for both chronic hepatitis B and C) | 24 weeks after treatment initiation
  Sustained virological response （Able to sustain an undetectable viral load for a period）
Serological responses(for chronic hepatitis B only) | 48 weeks after treatment initiation
  Hepatitis B e antigen (HBeAg) seroconversion(HBeAg loss and presence of anti-HBe) and hepatitis B surface antigen(HBsAg) seroconversion (HBsAg loss and presence of anti-HBs)

SECONDARY OUTCOMES:
Histological responses(for both chronic hepatitis B and C) | 48 weeks after treatment initiation
  Significant improvement in fibrosis was defined as a decrease in the Ishak score of at least 1 point; (the Ishak score describes six stages of fibrosis, 0 for No fibrosis and 6 for Cirrhosis; higher the Ishak score is, more severe the fibrosis is).

CONTACTS AND LOCATIONS:
Overall Officials: Wenhong Zhang, Professor, Study Chair — Huashan Hospital
Locations (1):
- Huashan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Maucort-Boulch D, de Martel C, Franceschi S, Plummer M. Fraction and incidence of liver cancer attributable to hepatitis B and C viruses worldwide. Int J Cancer. 2018 Jun 15;142(12):2471-2477. doi: 10.1002/ijc.31280. Epub 2018 Feb 9. PMID 29388206
- [Background] Polaris Observatory Collaborators. Global prevalence, treatment, and prevention of hepatitis B virus infection in 2016: a modelling study. Lancet Gastroenterol Hepatol. 2018 Jun;3(6):383-403. doi: 10.1016/S2468-1253(18)30056-6. Epub 2018 Mar 27. PMID 29599078